CLINICAL TRIAL: NCT00563979
Title: Enhancement of Macular Pigment Density by Oral Lutein Supplementation
Acronym: EMPOLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Sebastian Wolf, Director, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KEK 152/07
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Age-Related Maculopathies
Keywords: age related macular degeneration; supplementation; macular pigment
MeSH Terms: conditions — Macular Degeneration | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): VitaluxPlus®
  Interventions: Dietary Supplement: VitaluxPlus®
- 2 (Active Comparator): Omega 3
  Interventions: Dietary Supplement: Omega 3

INTERVENTIONS:
Dietary Supplement: VitaluxPlus® — 1 tablet daily
  Arms: 1
Dietary Supplement: Omega 3 — 1 tablet daily
  Arms: 2

SUMMARY:
The primary objective of EMPOLS is an increase in macular pigment density (MPD) and contrast sensitivity (CS) after six months supplementation of oral non-compound ester Lutein 10 mg daily, contained in VitaluxPlus®.

DETAILED DESCRIPTION:
The primary objective of EMPOLS is an increase in macular pigment density (MPD) and contrast sensitivity (CS) after six months supplementation of oral non-compound ester Lutein 10 mg daily, contained in VitaluxPlus®. Primary variable for a significant change will be 10% increase compared to baseline MPD.

The measurement will be carried out by means of a modified confocal scanning laser ophthalmoscope (HRA) recording autofluorescence images at 488 nm and 514 nm 6. MPD is determined on MPD maps within 0.5 degrees around the center of the fovea. All MPD measurements and photographs will by performed by the Bern Photographic Reading Center (BPRC). Complete examination of study patients comprises testing of standardized visual acuity (ETDRS-VA), visual contrast sensitivity (CS), biomicroscopy, fundus photography, and a blood sample. Participating patients also have to fill out a food frequency questionnaire (FFQ-Bern) allowing for correction of additional lutein intake by regular diet. Moreover possible confounding factors e.g. as sunlight exposure or smoking habits will be assessed. Secondary objective of EMPOLS is the effect of oral non-compound ester lutein supplementation on CS and ETDRS-VA during one year. The variable for a significant change in ETDRS-VA is loss or gain of 7 letters on the ETDRS chart, for a change in CS: loss or gain of at least four letters on the Pelli-Robson CS Chart. Additionally, serum carotenoid levels of lutein will be determined by high performance liquid chromatography (HPLC) for each visit 1.

ELIGIBILITY:
Inclusion Criteria:

* age related maculopathy

Exclusion Criteria:

* exudative age related degeneration

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Macular pigment density | 6 months

SECONDARY OUTCOMES:
contrast sensitivity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolf, MD, Study Director — University of Bern; Ute Wolf-Schnurrbusch, MD, Principal Investigator — University of Bern
Locations (1):
- Klinik und Poliklinik für Augenheilkunde, University Bern, Bern, Switzerland

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300
- [Derived] Wolf-Schnurrbusch UE, Zinkernagel MS, Munk MR, Ebneter A, Wolf S. Oral Lutein Supplementation Enhances Macular Pigment Density and Contrast Sensitivity but Not in Combination With Polyunsaturated Fatty Acids. Invest Ophthalmol Vis Sci. 2015 Dec;56(13):8069-74. doi: 10.1167/iovs.15-17586. PMID 26720458